CLINICAL TRIAL: NCT03860597
Title: Memantine Effects on Sensorimotor Gating and Neurocognition in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Neal R. Swerdlow, M.D., Ph.D., Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01MH094320 (NIH)
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Schizoaffective Disorder; Healthy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Memantine (Active Comparator)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Memantine — To assess the acute effects of MEM (0 vs. 20 mg) on measures of auditory processing fidelity, auditory learning and EAIP, in AP-medicated adult SZ patients and HS.
  Arms: Memantine
Drug: Placebos — To assess the acute effects of MEM (0 vs. 20 mg) on measures of auditory processing fidelity, auditory learning and EAIP, in AP-medicated adult SZ patients and HS.
  Arms: Placebo

SUMMARY:
This application seeks to determine if neurophysiological metrics of memantine (MEM)-enhanced early auditory information processing (EAIP) in schizophrenia (SZ) mediate gains in auditory processing fidelity (APF) and auditory learning.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia OR schizoaffective-depressed OR healthy subjects
* ages 18-50 for all subjects
* double barrier contraception for all subjects
* not pregnant for all subjects

Exclusion Criteria:

* DSM-IV Axis I or II Diagnosis for for healthy subjects
* MEM or amantadine for patients
* current substance abuse for all subjects
* current recreational drug use for all subjects
* history of other significant medical illness (e.g. cancer, diabetes, heart disease, HIV, seizures) for all subjects
* open head injury or closed head injury with loss of consciousness > 1 min for all subjects
* hearing or visual impairment for all subjects
* pregnancy for all subjects
* dementia for all subjects
* mental retardation for all subjects

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Teaching Facility (CTF-B102) at UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Molina JL, Voytek B, Thomas ML, Joshi YB, Bhakta SG, Talledo JA, Swerdlow NR, Light GA. Memantine Effects on Electroencephalographic Measures of Putative Excitatory/Inhibitory Balance in Schizophrenia. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Jun;5(6):562-568. doi: 10.1016/j.bpsc.2020.02.004. Epub 2020 Feb 22. PMID 32340927

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine; Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo; Healthy Subjects: Placebo 1st, Then 20 mg Memantine; Healthy Subjects: 20 mg Memantine 1st, Then Placebo: Memantine: To assess the acute effects of MEM (0 vs. 20 mg) on measures of auditory processing fidelity, auditory learning and EAIP, in AP-medicated adult SZ patients and HS.
  Placebos: To assess the acute effects of MEM (0 vs. 20 mg) on measures of auditory processing fidelity, auditory learning and EAIP, in AP-medicated adult SZ patients and HS.
Period: Overall Study
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Started | 11 | 11 | 10 | 10
Completed | 11 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: 20 mg Memantine 1st, Then Placebo | Total
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 10 | 10 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 40.1 [26 to 54] | 41.0 [32 to 54] | 29.6 [18 to 49] | 29.3 [18 to 48] | 35.3 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 6 | 6 | 23
  Male | 5 | 6 | 4 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6 | 6 | 18
  Not Hispanic or Latino | 8 | 7 | 4 | 4 | 23
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 4 | 2 | 8
  Asian | 1 | 1 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 2 | 0 | 1 | 5
  White | 4 | 3 | 3 | 4 | 14
  More than one race | 1 | 3 | 0 | 1 | 5
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Prepulse Inhibition (PPI)
Description: PPI of the startle reflex is the automatic reduction in startle magnitude (assessed by EMG of orbicularis oculi) when a startling stimulus (40 ms 118 dB(A) noise burst; "PULSE") is preceded (10-120 msec) by a weak stimulus (here a 20 msec burst 16 dB over background "PREPULSE"). A %PPI metric is calculated based on the relative startle magnitude on (PREPULSE + PULSE) trials vs. PULSE alone trials. Possible maximal inhibition is 100%; there is no maximal "negative" value of inhibition. There is no clear "advantage" or "disadvantage" for lower or higher %PPI values, though on average, schizophrenia patients demonstrate lower % values compared to matched healthy subjects. Day 1 was baseline testing: testing occurred, data was collected, but no "intervention" was given. There were two possible "interventions": active (MEM 20 mg po) and placebo. One intervention was given on day 7 post baseline, the other intervention was given on day 14 post baseline, with order of intervention balanced.
Time Frame: 7 and 14 days post baseline
Measure: Mean (Standard Error); unit: % inhibition of startle
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Number analyzed (Participants) | 9 | 7 | 10 | 10
% inhibition of startle
  Placebo | 32.45 (5.11) | 26.85 (6.77) | 14.11 (8.97) | 11.78 (8.73)
  Memantine | 10.11 (12.88) | 20.55 (4.07) | 21.36 (4.56) | 25.55 (6.37)

2. Primary Outcome: Mismatch Negativity (MMN); Unit of Measure of MMN is Microvolts.
Description: 85 dB SPL stimuli were presented via Etymotic ER3-A insert earphones. A 4-tone auditory oddball paradigm with 82% standards & 18% deviant stimuli, differed from standard in pitch, duration, or both. A pseudorandomized sequence produced a minimum of 3 standard tones between each deviant stimulus. All tones had 5-ms rise/fall times presented with a fixed 500-ms stimulus onset asynchrony. Subjects viewed a silent movie & instructed to ignore auditory stimuli. EEG were continuously recorded at a sampling rate of 2048-Hz from 64 channels, using BioSemi ActiveTwo system & downsampled to 512-Hz. Deviant-minus-standard difference waves were generated for each deviant type & low-pass filtered (20-Hz zerophase shift, 24 dB/octave rolloff). MMN was computed as mean amplitude across 135-205 ms range for each deviant type in difference waveforms at electrode Fz. Data were analyzed by RM-ANOVA, with diagnosis as a between-subject factor, & drug condition (placebo vs MEM) as a within-subject factor.
Time Frame: 7 and 14 days post baseline
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Number analyzed (Participants) | 11 | 10 | 9 | 9
microvolts
  Placebo | -3.15 (0.45) | -1.60 (0.31) | -3.52 (0.50) | -3.52 (0.50)
  Memantine | -2.44 (0.54) | -1.70 (0.28) | -3.28 (0.50) | -3.28 (0.50)

3. Primary Outcome: Gamma Auditory Steady-state Response (ASSR). The Primary Unit of Measure of Auditory Steady State Response (ASSR) is Gamma Evoked Power (γEP), Expressed as "Microvolts-squared".
Description: 1 ms, 85 dB clicks were presented in 500 ms trains at a frequency of 40 Hz; 250 click trains were played (inter-train interval=0.5 s). EEG was continuously recorded with 64-channel BioSemi ActiveTwo system (sampling rate=2048 Hz). Data processed offline via Matlab, EEGlab, & BrainVision Analyzer. Continuous data were segmented relative to stimulus onset (-100 ms to 500 ms) & each epoch was baseline-corrected relative to 100 ms pre-stimulus interval. γEP was assessed based on first 100 artifact-free epochs at Fz. Averaged epochs across click trains were transformed into power spectrum via fast Fourier transform using a bin width of 2 Hz. 40 Hz power spectrum was averaged across 4 Hz band from 38-42 Hz. Data were analyzed by RM-ANOVA, with diagnosis as a between- & drug condition (placebo vs MEM) as a within-subject factor. Analyses revealed robust & time bin-independent effects of diagnosis & drug across 200-500 ms window & thus this interval was the focus of all subsequent analyses.
Time Frame: 7 and 14 days post baseline
Measure: Mean (Standard Error); unit: Microvolts-squared
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Number analyzed (Participants) | 11 | 10 | 9 | 9
Microvolts-squared
  Placebo | 0.08 (0.02) | 0.07 (0.02) | 0.14 (0.03) | 0.14 (0.03)
  Memantine | 0.09 (0.04) | 0.06 (0.02) | 0.23 (0.06) | 0.23 (0.06)

ADVERSE EVENTS:
Time Frame: approximately 14 days
Description: Participants received their "interventions" twice: once on day 7 and once on day 14 post baseline. The the Frame of Adverse Events is the duration of time over which each participant was assessed, and this duration is 2 days: one day on day 7 pos baseline, plus a second day on day 14 post baseline.
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT03860597/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT03860597/SAP_001.pdf